CLINICAL TRIAL: NCT05179603
Title: Phase 2 Non-randomized, Open-label, Multi-cohort, Multicenter Study Assessing the Clinical Benefit of SAR444245 (THOR-707) With or Without Other Anticancer Therapies for the Treatment of Adults and Adolescents With Relapsed or Refractory B Cell Lymphoma
Brief Title: A Study of SAR444245 With or Without Other Anticancer Therapies for the Treatment of Adults and Adolescents With Relapsed or Refractory B Cell Lymphoma (Master Protocol) [Pegathor Lymphoma 205]
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early discontinuation based on strategic sponsor decision not driven by any safety concerns
Sponsor: Sanofi (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACT16941; U1111-1251-5834 (Registry Identifier: ICTRP); MK-3475-C39 (Other: Merck Sharp & Dohme LLC.); KEYNOTE-C39 (Other: Merck Sharp & Dohme LLC.); 2021-002150-91 (EudraCT Number)
Record Dates: First submitted 2021-12-16; First posted 2022-01-05 (Actual); Results first posted 2025-10-02 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Classic Hodgkin Lymphoma; Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — pembrolizumab; Drugs, Generic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort A: Pegenzileukin 24 μg/kg + Pembrolizumab (Experimental): Participants with classic Hodgkin lymphoma (cHL) who were anti-programmed cell death-ligand 1 (PD-L1)-naïve and had received at least 2 or 3 lines of systemic therapy received pegenzileukin 24 microgram per kilogram (μg/kg) via intravenous (IV) infusion over 30 minutes on Day 1 of each cycle (each cycle is 21 days), along with pembrolizumab 200 milligram (mg) via 30 minutes IV infusion on Day 1 of each 3-week treatment cycle (each cycle is 21 days) as third-line or fourth-line (3/4L) therapy, until disease progression (PD), unacceptable adverse event (AE) or other full permanent discontinuation criteria was met or completion of Cycle 35.
  Interventions: Drug: THOR-707; Drug: Pembrolizumab
- Cohort C1: (sub study 03) diffuse large B Cell lymphoma (DLBCL) (Experimental): Pegenzileukin administered every 2 weeks on Day 1 of each cycle (14 days per cycle) for up to 52 cycles.
  Interventions: Drug: THOR-707

INTERVENTIONS:
Drug: THOR-707 — Pharmaceutical Form: Solution for infusion Route of Administration: Intravenous infusion
  Other Names: Pegenzileukin
Drug: Pembrolizumab — Pharmaceutical Form: Solution for infusion Route of Administration: Intravenous infusion
  Other Names: KEYTRUDA® or generic
  Arms: Cohort A: Pegenzileukin 24 μg/kg + Pembrolizumab

SUMMARY:
This is a phase 2 multi-cohort, un-controlled, non-randomized, open-label, multi-center study that assessed the antitumor activity and safety of non-alpha interleukin (IL-2) SAR444245 with or without other anticancer therapies in participants aged 12 years and older with relapsed or refractory B cell lymphoma. This study was structured as a master protocol with separate sub studies designed to investigate the use of SAR444245 either with or without other anticancer therapies for the treatment of relapsed or refractory B cell lymphoma.

Substudy 1-Cohort A aimed to establish safety and preliminary anti-tumor activity for non-alpha interleukin (IL-2) SAR444245 combined with the anti-PD1 antibody, pembrolizumab in trial participants with classic Hodgkin lymphoma (cHL) who are anti-PD-(L)1-naive and have received at least 2 or 3 lines of systemic therapy.

Substudy 3-Cohort C1 aims to establish safety and preliminary anti-tumor activity for SAR444245 as monotherapy in trial participants with diffuse large B-cell lymphoma (DLBCL). Trial participants in this study must have received at least 2 lines of systemic therapy and have either stable or progressive disease 1-3 months post Health Authority approved Chimeric Antigen Receptor T-cell (CAR-T) treatment when given as last systemic treatment prior to study enrollment.

DETAILED DESCRIPTION:
The duration of the study for an individual participant started from the signature of the main informed consent and included:

a screening period of up to 28 days;

a treatment period [max] 35 cycles (21 days per cycle) for Cohort A and 52 cycles (14 days per cycle) for Cohort C1 or until occurrence of unacceptable toxicities or until PD;

an end-of-treatment visit at least approximately 30 days following the last administration of study drug (or until the participant receives another anticancer therapy, whichever is earlier);

and a follow-up visits 3 months after treatment discontinuation and every 3 months thereafter following, until disease progression, or initiation of another antitumor treatment, or death, whichever is earlier.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have been ≥ 12 years of age, at the time of signing the informed consent
* Disease location was amenable to tumor biopsy at baseline
* All participants must have had a measurable disease
* Both male and female participants agreed to use approved contraception methods; not pregnant or breastfeeding for female participants; no donation or cryopreservation of eggs (ova, oocytes) for female participants and sperms for male participants.
* Had to be capable of giving signed informed consent

For cohort A: Histologically or cytologically confirmed diagnosis of classic Hodgkin lymphoma (cHL), must have received at least two prior lines of systemic therapy for cHL, including at least one containing an anthracycline or brentuximab.

For cohort C1: Histologically confirmed diagnosis of diffuse large B Cell lymphoma (DLBCL), must have received at least two prior lines of systemic therapy for DLBCL, including one containing a combination of anthracycline and rituximab (or another anti-CD20 agent), with the last line of therapy a Health Authority approved CD19-directed CAR-T therapy. Patients must have BOR (Best Overall Response) of stable disease (SD) or progressive disease (PD) after CD-19 directed CAR-T therapy.

Exclusion Criteria:

Participants were excluded from the study if any of the following criteria applied:

* Eastern Cooperative Oncology Group (ECOG) performance status of ≥ 2 (≥ 16 years old). Lansky Scale (< 16 years old) ≤ 60%
* Poor bone marrow reserve
* Poor organ function
* Participants with baseline oxygen saturation (SpO2) ≤ 92% (without oxygen therapy)
* Lymphomatous involvement of the central nervous system
* History of allogenic or solid organ transplant
* Prior IV or subcutaneous anticancer therapy, investigational agent, major surgery within 21 days prior to initiation of IMP; oral anticancer therapy within 5 half-lives or completed palliative radiotherapy within 21 days prior to initiation of IMP
* Has received prior IL-2-based anticancer treatment
* Comorbidity requiring corticosteroid therapy
* Antibiotic use (excluding topical antibiotics) ≤ 14 days prior to first dose of IMP
* Severe or unstable cardiac condition within 6 months prior to starting study treatment
* Had active, known, or suspected autoimmune disease that has required systemic treatment in the past 2 years-Known second malignancy either progressing or requiring active treatment within the last 3 years
* Receipt of a live or live attenuated virus vaccination within 28 days of planned treatment start. Seasonal flu vaccines or SARS-CoV-2 vaccine that do not contain live virus were permitted

The above information is not intended to contain all considerations relevant to the potential participation in a clinical trial.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2024-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (8):
- Investigational Site Number : 0320005, CABA, Buenos Aires, Argentina
- Chile (4):
  - Investigational Site Number : 1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520004, Viña del Mar, Región de Valparaíso
  - Investigational Site Number : 1520001, Temuco
- Spain (3):
  - Investigational Site Number : 7240002, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240001, L'Hospitalet de Llobregat, Barcelona [Barcelona]
  - Investigational Site Number : 7240004, Madrid / Madrid, Madrid, Comunidad de

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: ACT16941 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25205&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 7 centers (corresponds to number of sites which screened at least one participant) in 3 countries from 07 December 2021 to 26 October 2022. Out of 19 participants who were screened, 14 participants were enrolled in the study.
Pre-assignment Details: The study was terminated based on strategic sponsor decision not driven by any safety concerns. The Cohort C1 was not initiated and no participants were enrolled.
  Note: Reason for not completed = Reason for permanent full intervention discontinuation.
Period: Overall Study
Arm/Group | Cohort A: Pegenzileukin 24 μg/kg + Pembrolizumab
Started | 14
Completed | 2
Not Completed | 12
Not completed — Unspecified: Not related to Coronavirus Disease 2019 (COVID-19) | 3
Not completed — Withdrawal by Subject | 1
Not completed — Progressive disease | 4
Not completed — Adverse event: Not related to COVID-19 | 4

BASELINE CHARACTERISTICS:
Population: The exposed population consisted of all participants who had given their informed consent and received at least one dose of study treatment.
Groups:
- Cohort A: Pegenzileukin 24 μg/kg + Pembrolizumab: Participants with cHL who were anti-PD-L1-naïve and had received at least 2 or 3 lines of systemic therapy received pegenzileukin 24 μg/kg via IV infusion over 30 minutes on Day 1 of each cycle (each cycle is 21 days), along with pembrolizumab 200 mg via 30 minutes IV infusion on Day 1 of each 3-week treatment cycle (each cycle is 21 days) as 3/4L therapy, until PD, unacceptable AE or other full permanent discontinuation criteria was met or completion of Cycle 35.
Arm/Group | Cohort A: Pegenzileukin 24 μg/kg + Pembrolizumab
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.6 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate (CRR)
Description: The CRR was defined as the percentage of participants who had a complete response (CR) as the best overall response (BOR) as per Investigator assessment (Lugano response criteria 2014). The BOR was defined as the BOR observed from the date of first study treatment until PD, death, cut-off date or initiation of subsequent anti-cancer therapy, whichever occurred first. CR based on computed tomography (CT)-based response: lymph nodes and extralymphatic sites with target nodes/nodal masses must regress to <=1.5 centimeter (cm) in longest transverse diameter of a lesion (LDi) and no extralymphatic sites of disease.
Time Frame: From first dose of study treatment administration (Day 1) up to approximately 21 months
Population: The efficacy population consisted of all participants from the exposed population with at least one evaluable post-baseline tumor assessment or who permanently discontinued study treatment.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Pegenzileukin 24 μg/kg + Pembrolizumab
Number analyzed (Participants) | 14
percentage of participants | 71.4 [46.0 to 89.6]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of the participants with CR or partial response (PR) as the BOR as per Investigator assessment (Lugano response criteria 2014). The BOR was defined as the BOR observed from the date of first study treatment until PD, death, cut-off date or initiation of subsequent anti-cancer therapy, whichever occurs first. CR (CT-based response): lymph nodes and extralymphatic sites with target nodes/nodal masses must regress to <=1.5cm in LDi and no extralymphatic sites of disease. PR (CT-based response): lymph nodes and extralymphatic sites with >=50% decrease in sum of the product of the perpendicular diameters for multiple lesions (SPD) of upto 6 target measurable nodes and extranodal sites. A lesion too small to measure on CT, 5 millimeter (mm) X 5mm used as default value. No longer visible, 0 X 0 mm. A node >5mm X 5mm, but smaller than normal, actual measurement used.
Time Frame: From first dose of study treatment administration (Day 1) up to maximum exposure of study treatment; approximately 28 months
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Pegenzileukin 24 μg/kg + Pembrolizumab
Number analyzed (Participants) | 14
percentage of participants | 92.9 [70.3 to 99.6]

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An SAE was any AE that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or was an important medical event. TEAEs were defined as AEs that developed, worsened (according to the Investigator's opinion) or became serious during the TE period.
Time Frame: From first dose of study treatment (Day 1) up to 30 days after the last dose of study treatment; approximately 29 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Pegenzileukin 24 μg/kg + Pembrolizumab
Number analyzed (Participants) | 14
Participants
  TEAEs | 14
  TESAEs | 5

4. Secondary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: Selected events that occurred during the DLT observation period were considered as DLT unless due to PD or to a cause obviously unrelated to pegenzileukin. Selected events included: grade 4 neutropenic fever, grade 4 thrombocytopenia associated with clinically significant bleeding that required clinical intervention, grade 3 or above alanine aminotransferase or aspartate aminotransferase in combination with a bilirubin >2 × upper limit of normal with no evidence of cholestasis or another cause, such as viral infection or other drugs, grade 3 or above vascular leak syndrome, grade 3 or above hypotension, grade 3 or above cytokine release syndrome, grade 3 or above AE that did not resolve to grade <=2 within 7 days of starting accepted standard of care medical management.
Time Frame: From Day 1 to Day 21 of Cycle 1 (each cycle is 21 days)
Population: DLT-evaluable population consisted of all exposed participants in safety run-in part who had been treated and observed for DLT observation period. Any participants who had experienced a DLT during DLT observation period were also DLT-evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Pegenzileukin 24 μg/kg + Pembrolizumab
Number analyzed (Participants) | 7
Participants | 1

5. Secondary Outcome: Time to Response (TTR)
Description: The TTR was defined as the time from the first administration of study treatment to the first tumor assessment at which the overall response was recorded as PR or CR determined by Investigator (Lugano response criteria 2014). CR (CT-based response): lymph nodes and extralymphatic sites with target nodes/nodal masses must regress to <=1.5cm in LDi and no extralymphatic sites of disease. PR (CT-based response): lymph nodes and extralymphatic sites with >=50% decrease in sum of the product of the perpendicular diameters for multiple lesions (SPD) of upto 6 target measurable nodes and extranodal sites. A lesion too small to measure on CT, 5 millimeter (mm) X 5mm used as default value. No longer visible, 0 X 0 mm. A node >5mm X 5mm, but smaller than normal, actual measurement used.
Time Frame: as for outcome 2
Population: The efficacy population consisted of all participants from the exposed population with at least one evaluable post-baseline tumor assessment or who permanently discontinued study treatment. Only participants with confirmed CR or PR were analyzed.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort A: Pegenzileukin 24 μg/kg + Pembrolizumab
Number analyzed (Participants) | 13
months | 2.0 [2 to 2]

6. Secondary Outcome: Duration of Response (DoR)
Description: The DoR was defined as the time from the first tumor assessment at which the overall response was recorded as PR or CR until PD determined by Investigator (Lugano response criteria 2014), or death from any cause, whichever occurred first. CR (CT-based response): lymph nodes and extralymphatic sites with target nodes/nodal masses must regress to <=1.5cm in LDi and no extralymphatic sites of disease. PR (CT-based response): lymph nodes and extralymphatic sites with >=50% decrease in sum of the product of the perpendicular diameters for multiple lesions (SPD) of upto 6 target measurable nodes and extranodal sites. A lesion too small to measure on CT, 5 millimeter (mm) X 5mm used as default value. No longer visible, 0 X 0 mm. A node >5mm X 5mm, but smaller than normal, actual measurement used.
Time Frame: as for outcome 2
Population: as for outcome 5
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Cohort A: Pegenzileukin 24 μg/kg + Pembrolizumab
Number analyzed (Participants) | 13
months | NA [6.3 to NA] — NA indicates that the median and upper limit of 90% confidence interval (CI) were not estimable due to insufficient number of participants with events.

7. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR was defined as percentage of participants with clinical benefit (CR or PR as BOR, or stable disease [SD] lasting at least 6 months) determined by Investigator per Lugano response criteria 2014. BOR was defined as BOR observed from date of first study treatment until PD, death, cut-off date or initiation of subsequent anti-cancer therapy, whichever occurred first. CR (CT-based response): lymph nodes and extralymphatic sites with target nodes/nodal masses must regress to <=1.5cm in LDi and no extralymphatic sites of disease. PR (CT-based response): lymph nodes and extralymphatic sites with >=50% decrease in SPD of upto 6 target measurable nodes and extranodal sites. A lesion too small to measure on CT, 5mm X 5mm used as default value. No longer visible, 0 X 0 mm. A node >5mm X 5mm, but smaller than normal, actual measurement used. SD (CT-based response): <50% decrease from baseline in SPD of up to 6 dominant, measurable nodes and extranodal sites; no criteria for PD met.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Pegenzileukin 24 μg/kg + Pembrolizumab
Number analyzed (Participants) | 14
percentage of participants | 92.9 [70.3 to 99.6]

8. Secondary Outcome: Progression Free Survival (PFS)
Description: The PFS was defined as the time from the date of first study treatment administration to the date of the first documented PD determined by Investigator (Lugano response criteria 2014), or death due to any cause. PFS (CT-based response): An individual node/lesion had to be abnormal with: LDi >1.5 cm and increased by >=50% from positron emission tomography nadir and an increase in LDi or shortest axis perpendicular to the LDi from nadir, 0.5cm for lesions <=2 cm, 1.0cm for lesions>2 cm. In the setting of splenomegaly, the splenic length must be increased by >50% of the extent of its prior increase beyond baseline. If there was no prior splenomegaly, increase by at least 2 cm from baseline. For new lesions regrowth of previously resolved lesions: a new node >1.5 cm in any axis, a new extranodal site>1.0 cm in any axis.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Cohort A: Pegenzileukin 24 μg/kg + Pembrolizumab
Number analyzed (Participants) | 14
months | NA [8.3 to NA] — NA indicates that the median and upper limit of 90% CI were not estimable due to insufficient number of participants with events.

9. Secondary Outcome: Plasma Concentrations of Pegenzileukin
Description: Blood samples were collected at specified timepoints for the assessment of plasma concentrations of pegenzileukin .
Time Frame: Cycle 1 Day 2, Cycle 1 Day 3 (each cycle is 21 days)
Population: The pharmacokinetic (PK) population consisted of all participants from the exposed population with at least one PK concentration available after the first dose of study treatment. Only participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Cohort A: Pegenzileukin 24 μg/kg + Pembrolizumab
Number analyzed (Participants) | 9
nanogram/milliliter (ng/mL)
  Cycle 1 Day 2 | 191.7 (78.4)
  Cycle 1 Day 3: number analyzed (Participants) | 8
  Cycle 1 Day 3 | 95.2 (75.8)

10. Secondary Outcome: Concentration at End of Infusion (Ceoi) of Pegenzileukin
Description: Blood samples were collected at specified timepoints for the assessment of Ceoi of pegenzileukin .
Time Frame: Cycles 1, 2, 4, 7, 10, 15 (each cycle is 21 days)
Population: The PK population consisted of all participants from the exposed population with at least one PK concentration available after the first dose of study treatment. Only participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort A: Pegenzileukin 24 μg/kg + Pembrolizumab
Number analyzed (Participants) | 13
ng/mL
  Cycle 1 | 438.2 (238.6)
  Cycle 2: number analyzed (Participants) | 9
  Cycle 2 | 405.4 (255.6)
  Cycle 4: number analyzed (Participants) | 6
  Cycle 4 | 435.2 (173.9)
  Cycle 7: number analyzed (Participants) | 6
  Cycle 7 | 594.7 (208.4)
  Cycle 10: number analyzed (Participants) | 4
  Cycle 10 | 596.3 (181.3)
  Cycle 15: number analyzed (Participants) | 1
  Cycle 15 | 325.0 (NA) — NA indicates that the standard deviation (SD) was not estimable for 1 participant.

11. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADA) Against Pegenzileukin
Description: Blood samples were collected at specified timepoints to assess the presence of ADA against pegenzileukin . Treatment-emergent ADA was defined as at least one treatment-induced or treatment-boosted ADA. Treatment-induced ADA was defined as ADA that developed during the TE period and without pre-existing ADA (including participants without pre-treatment samples). Treatment-boosted ADA was defined as pre-existing ADA that was boosted during the TE period to a significant higher titer than the baseline. Number of participants with treatment-emergent ADA is presented.
Time Frame: as for outcome 3
Population: ADA population consisted of all participants from exposed population with at least one ADA result (positive, negative or inconclusive) after the first dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Pegenzileukin 24 μg/kg + Pembrolizumab
Number analyzed (Participants) | 12
Participants | 3

ADVERSE EVENTS:
Time Frame: Adverse events data was collected from first dose of study treatment (Day 1) up to 30 days after the last dose of study treatment, approximately 29 months. All-cause mortality (death) was assessed from first dose of study treatment (Day 1) up to end of follow-up for each participant, approximately 32 months.
Description: Analysis was performed on the exposed population.
Arm/Group | Cohort A: Pegenzileukin 24 μg/kg + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 5/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Pegenzileukin 24 μg/kg + Pembrolizumab (N=14)
Septic Shock (Infections and infestations) | 1 (2)
Urinary Tract Infection Fungal (Infections and infestations) | 1 (1)
Cytokine Release Syndrome (Immune system disorders) | 3 (4)
Hypophysitis (Endocrine disorders) | 1 (1)
Immune-Mediated Hypophysitis (Endocrine disorders) | 1 (1)
Immune-Mediated Myocarditis (Cardiac disorders) | 2 (2)
Immune-Mediated Hepatitis (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Pegenzileukin 24 μg/kg + Pembrolizumab (N=14)
Bronchitis (Infections and infestations) | 1 (1)
Dengue Fever (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2)
Oral Herpes (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Respiratory Tract Infection Viral (Infections and infestations) | 2 (2)
Rhinitis (Infections and infestations) | 1 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (2)
Urinary Tract Infection (Infections and infestations) | 2 (6)
Viral Parotitis (Infections and infestations) | 1 (1)
Viral Pharyngitis (Infections and infestations) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Cytokine Release Syndrome (Immune system disorders) | 1 (1)
Glucocorticoid Deficiency (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 3 (3)
Immune-Mediated Hypothyroidism (Endocrine disorders) | 1 (1)
Thyroiditis (Endocrine disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (3)
Neuralgia (Nervous system disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Vitreous Floaters (Eye disorders) | 1 (1)
Vasculitis (Vascular disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (3)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 3 (4)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1 (1)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 2 (4)
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Vitiligo (Skin and subcutaneous tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Pyrexia (General disorders) | 3 (3)
Swelling Face (General disorders) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 1 (1)
Blood Alkaline Phosphatase Increased (Investigations) | 1 (2)
Blood Bilirubin Increased (Investigations) | 1 (1)
Blood Sodium Decreased (Investigations) | 1 (1)
Blood Thyroid Stimulating Hormone Increased (Investigations) | 1 (1)
Lymphocyte Count Increased (Investigations) | 1 (1)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 11 (94)

LIMITATIONS AND CAVEATS:
The study was terminated based on strategic sponsor decision not driven by any safety concerns and no participants were enrolled in Cohort C1.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/03/NCT05179603/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/03/NCT05179603/SAP_001.pdf